CLINICAL TRIAL: NCT01191164
Title: A Prospective Study to Evaluate the Feasibility of Partial Breast Irradiation Utilizing Permanent Breast Seed Implant in British Columbia
Brief Title: Pilot Study of Partial Breast Irradiation Utilizing Permanent Breast Seed Implant to Treat Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCCA-H09-01053
Record Dates: First submitted 2010-08-25; First posted 2010-08-30 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Brachytherapy, Partial Breast Irradiation, Breast Seed Implant, Palladium Seeds
MeSH Terms: conditions — Breast Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Arm (Experimental)
  Interventions: Procedure: Partial Breast Irradiation Utilizing Permanent Breast Seed Implant

INTERVENTIONS:
Procedure: Partial Breast Irradiation Utilizing Permanent Breast Seed Implant — Target Volumes: The surgical cavity will be assessed with US & CT scans. The Clinical Target Volume (CTV) will encompass the surgical cavity plus 1 cm uniform expansion. The Planning Target Volume (PTV) will be the CTV plus 0.5 cm.
  Dose Selection/Prescription: A minimal peripheral dose of 90 Gy (same as in the OCC study) will be prescribed to the PTV. This dose is chosen as biologically equivalent, over a 2 month period, to 50Gy in 25 fractions, for α/β of 2Gy54.
  Implant Procedure and QA: This will be performed as an outpatient procedure under conscious sedation and local anesthesia, by a team with several years experience in brachytherapy and conscious sedation administration. The technique used in this pilot study will be based on the OCC technique. It is intended that two oncologists and one physicist will spend 2-3 days at the OCC to acquire detailed and firsthand knowledge of the technique and its implementation at that centre.
  Other Names: Brachytherapy

SUMMARY:
Background: Recent single arm studies have suggested that partial breast irradiation (PBI), delivered in a relatively short overall treatment time of a few days, may be an effective alternative to adjuvant whole breast irradiation (WBI) delivered over a number of weeks. Several PBI modalities and techniques have been investigated, including interstitial brachytherapy and external beam radiation therapy, most often given over the course of one week of twice daily outpatient treatments. One randomized study has shown equivalency between WBI and PBI using brachytherapy. There are currently three large phase-III randomized studies comparing PBI to WBI.

Permanent Breast Seed Implant (PBSI) is the newest PBI technique which has been piloted at the Odette Cancer Centre (OCC) in Toronto. The main advantage of this technique is that it requires only one out-patient procedure. The treatment is administered by implanting radioactive Palladium (103Pd) seeds into the tumor bed region in a 1 to ½ hour outpatient procedure, after which the patient is discharged home to resume her normal living activities. This PBI procedure was shown to be well tolerated with minimal acute toxicity. Estimated partner radiation exposure was well within internationally acceptable levels. Subjects with a seroma >2cm were, however, excluded.

Hypothesis: PBSI is a feasible, safe, and acceptable treatment option for the subject and her partner in the context of medical practice and resources in BC.

Objectives: In subjects who have undergone breast conserving surgery for early breast cancer:

1. To determine the technical feasibility of PBSI in BC
2. To measure the subject's partner in terms of radiation protection
3. To evaluate acceptability of PBSI by the subject
4. To assess resource requirements for PBSI

Method: This is a single arm feasibility study. Five women who had undergone breast conserving surgery for breast cancer with low risk of local recurrence will be accrued. This study will adhere to a detailed written protocol for radiation measurements and protection.

Subjects will undergo PBSI within 4-14 weeks from last breast surgery. The procedure will be performed in an outpatient setting, under conscious sedation and local anesthesia, by a team with a wide brachytherapy experience. The technique used in this feasibility study will be based on the OCC technique. It is intended that two oncologists and one physicist will spend 2-3 days at the OCC to acquire detailed and firsthand knowledge of the technique as implemented at that centre.

The OCC technique is US-based; in this study, however, an additional CT-assisted planning component will be investigated building on the experience of the VIC team which conducted the BC Cancer Agency Vancouver Island Centre's pilot study of CT-based multi-catheter brachytherapy PBI.

Systemic therapy will be according to BCCA guidelines; however, subjects requiring adjuvant chemotherapy will be excluded from this study. Subjects will be followed prospectively for 5 years for evaluation of toxicity, QOL and cosmesis. Disease status will be recorded.

Relevance: Completing adjuvant breast irradiation with a single out-patient treatment could significantly improve QOL and convenience for patients choosing breast conserving therapy. Confirming the technical feasibility and safety of PBSI is needed before progressing to larger prospective evaluation of this novel adjuvant radiation therapy technique as a viable treatment option for women in British Columbia.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject with a pathologically-confirmed diagnosis of invasive ductal carcinoma.
2. Tumor size < 2cm.
3. Negative axillary node involvement, determined by either

   1. Sentinel node biopsy,
   2. Axillary node dissection removing > 6 nodes
4. No evidence of metastatic disease.
5. Treated by BCS with microscopically clear resection margins (> 2mm to ink) for invasive and non-invasive disease or no residual disease on re-excision.

Exclusion Criteria:

1. Age < 60 years.
2. Subjects who will receive adjuvant chemotherapy.
3. A known deleterious mutation in BRCA-1 and/or BRCA-2.
4. Extensive DCIS, mammographically or pathologically.
5. Tumor histology of pure lobular carcinoma (invasive or in-situ).
6. Adenoid cystic and non-epithelial malignancies (e.g. sarcoma or lymphoma).
7. Lymphovascular invasion (LVI) present.
8. Bilateral invasive malignancy of the breast (synchronous or metachronous).
9. More than one ipsilateral breast primary tumor.
10. Previous irradiation to the ipsilateral breast.
11. Presence of an ipsilateral breast implant.
12. Serious non-malignant disease that precludes radiation treatment or conscious sedation.
13. Unable for any reason to undergo PBSI within 14 weeks of the last breast surgery.
14. Concomitant malignancies, except non-melanoma skin cancer and carcinoma in situ of any site.
15. Significant persistent post-surgical complications.
16. Currently pregnant or lactating.
17. Psychiatric or addictive disorders which would preclude obtaining informed consent.
18. Subject not committed to at least 3 years of follow-up.
19. Low CBC levels: HB < 100 - Platelets < 100 - Neutrophil count < 1
20. Close partner not consenting
21. Inability to confidently localize/delineate the surgical cavity on CT and/or US.
22. Subject not suitable for a minimum 2-plane implant based on tumor location/breast size.
23. Seroma exceeding 3cm
24. Seroma within the inner quadrants

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Technical parameters of the implant | Measured once for each subject at a post-implant CT on the same day as the implant procedure. Will be assessed collectively once treatment is completed for all 5 subjects.
  Implant technical parameters will include:
  * SC (Surgical Cavity/Seroma) volume (average & range)
  * PTV (average & range)
  * Number of seeds per implant (average & range)
  * Average total seed activity per implant
  * From DVH, average and range of:
    * V90
    * V100
    * V150
    * V200
    * DHI
    * Number of seeds at a distance 5 mm or less from the skin surface
    * Absolute (cc) and proportional (%) volume of ipsilateral breast receiving 90%, 50% and 10 % of the prescribed dose
Seed motion at 1 month | Measured once for each subject at CT performed 1 month after implant procedure. Will be assessed collectively once treatment is completed for all 5 subjects.
  Seed motion at 1 month will be determined from CT performed one month after PBSI
Exposure Dose (ED) average and range for close partners | Once per week for 4 weeks following implant
  For the purpose of this study, the subject and her partner, if any, will be asked to wear a small, unobtrusive, radiation measuring device around one arm for a period of 4 weeks. The amount of radiation from the breast implant to the subject and partner (if any) will be measured once per week for 4 weeks, during which time the level of radiation from the breast will become so low that subject will no longer need to wear the patch.
Acute radiation toxicity | Prior to implant, and at 1, 4 & 12 weeks after implant.
  Acute Toxicity Assessment: Acute toxicity will be assessed by a clinical trial nurse or clinical research associate (CRA) using the NCI Common Toxicity Criteria for Adverse Events (NCI CTCAE), Version 3.0 (see Appendix V). Acute toxicity will be assessed prior to PBSI and 1, 4 & 12 weeks post-PBSI.
Adverse cosmetic outcome as a measure of late radiation morbidity | Before implant, at 1, 3 and 5 years post-implant.
  Late Radiation Toxicity Assessment: Late RT toxicity will be assessed by a clinical trial nurse or CRA using the relevant items from the RTOG/EORTC late RT toxicity scale58, subject-administered OCOG Cosmetic Module, EORTC Cosmetic Rating System, and Digital Photographs for Cosmetic Assessment.
Subject's Quality of Life | 2 weeks prior to the procedure and at 1, 4 & 12 weeks and 1, 3 & 5 years follow-up visits.
  Quality of Life Assessment: Quality of life will be assessed using the self administered EORTC Quality of Life QLQ C-30 Questionnaire within the 2 weeks prior to the procedure and at 1, 4 & 12 weeks and 1, 3 & 5 years follow-up visits.
Subject satisfaction | 1 and 12 weeks after implant
  Subject Satisfaction with the PBSI procedure: Subject satisfaction with the procedure will be assessed using a specifically designed questionnaire, administered at 1 and 12 weeks follow-up visits.

SECONDARY OUTCOMES:
Average human resource cost per a PBSI, including oncologists, physicists, therapists, and nursing time (time spent by different personnel on various treatment components). | After completion of implant procedure and 5 years of follow up.
Cost of seeds and consumables for each implant (and relationship to PTV). | After completion of implant procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hosam A Kader, MD, Principal Investigator — BCCA, Department of Radiation Oncology
Locations (1):
- British Columbia Cancer Agency, Victoria, British Columbia, Canada